CLINICAL TRIAL: NCT00005762
Title: Pharmacokinetic Interaction Studies of Amprenavir (APV), Efavirenz (EFV), and a Second Protease Inhibitor in HIV-Seronegative Volunteers
Brief Title: Drug Interactions of Amprenavir and Efavirenz, in Combination With a Second Protease Inhibitor, in HIV-Negative Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: A5043; 10671 (Registry Identifier: DAIDS ES); ACTG A5043
Record Dates: First submitted 2000-05-25; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Drug Interactions; Drug Therapy, Combination; HIV Protease Inhibitors; Ritonavir; Dosage Forms; Saquinavir; VX 478; Anti-HIV Agents; Nelfinavir; Pharmacokinetics; efavirenz
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Ritonavir; amprenavir; Nelfinavir; efavirenz; Saquinavir

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Ritonavir
Drug: Amprenavir
Drug: Nelfinavir mesylate
Drug: Efavirenz
Drug: Saquinavir

SUMMARY:
The purpose of this study is to measure the blood levels of amprenavir (APV) alone, APV combined with efavirenz (EFV), and APV/EFV combined with a third drug (nelfinavir [NFV], indinavir [IDV], ritonavir soft gel capsules [RTV sgc], or saquinavir soft gel capsules [SQV sgc]).

Anti-HIV therapy with 3 or 4 drugs is currently the recommended approach for treating HIV infections. Doctors need to know the best dosages of certain drugs when they are given in combination. This study will measure the blood levels of APV alone, APV combined with EFV, and APV/EFV plus a second PI in healthy volunteers. It will study the safety and tolerance of these drugs.

DETAILED DESCRIPTION:
Triple-drug antiretroviral regimens have become the recommended approach to therapy for HIV infection. [AS PER AMENDMENT 12/4/00: The clinical use of multiple-drug antiretroviral regimens containing various combinations of nucleoside reverse transcriptase inhibitors (NRTIs), nonnucleoside reverse transcriptase inhibitors (NNRTIs), and protease inhibitors (PIs) has become a widespread approach to therapy for HIV infection, especially for patients previously treated with PIs.] Since the introduction of PIs, a greater awareness of the relationship between optimal suppression of viral replication, genotypic resistance, and viral rebound has led to the design of more potent antiretroviral drug combinations. Two ACTG clinical trials addressing the issue of virologic failure utilize antiviral regimens that include 2 NRTIs, 2 PIs (one of which is APV), and EFV (NNRTI). Although this drug combination is logical, there is limited PK data to guide the dosing selection. This study enrolls healthy volunteers to obtain PK profiles and metabolic assessments of APV/EFV before and after the addition of a second PI [AS PER AMENDMENT 12/4/00: APV alone, APV combined with EFV, and APV/EFV combined with a second PI].

Upon study entry, volunteers receive APV plus EFV for 2 weeks. [AS PER AMENDMENT 12/4/00: Volunteers receive a single dose of APV alone on Day 0, EFV alone on Days 1 to 10, and APV combined with EFV on Days 11 to 13.] After 2 weeks [AS PER AMENDMENT 12/4/00: After completion of the second PK visit], volunteers are randomized to 1 of 5 treatment arms to add a second PI to the APV/EFV drug combination for 2 more weeks [AS PER AMENDMENT 12/4/00: for at least 1 week]. The treatment arms are as follows:

Arm A (control arm): APV and EFV alone. Arm B: APV and EFV plus IDV [AS PER AMENDMENT 12/4/00: APV and EFV plus NFV]. Arm C: APV and EFV plus NFV [AS PER AMENDMENT 12/4/00: APV and EFV plus IDV]. Arm D: APV and EFV plus RTV sgc. Arm E: APV and EFV plus SQV sgc. On Day 14, 15, or 16, volunteers return to the clinic for PK testing following the dual-drug regimen, and again on Day 29, 30, or 31 following the triple-drug regimen (or continued dual-drug regimen for Arm A). [AS PER AMENDMENT 12/4/00: Volunteers attend clinics for PK testing on Days 0 and 1 (first visit), after taking the dual-drug regimen for at least 3 days (second visit, e.g., on Day 14 or after), and after taking the triple-drug regimen (or, if in Arm A, after continuing on the dual-drug regimen) for at least 7 days (third visit).] Before each PK testing, volunteers complete an Adherence Questionnaire. [AS PER AMENDMENT 12/4/00: The Adherence Questionnaire is administered at the second and third PK visits.] Volunteers maintain a food diary. Two to three weeks after completing the drug regimen [AS PER AMENDMENT 12/4/00: Within 2-3 weeks after the third PK visit], volunteers return to the clinic for evaluations and urine and blood sampling.

ELIGIBILITY:
Inclusion Criteria

Volunteers may be eligible for this trial if they:

* Are HIV negative.
* Are 18 to 65 years old.
* Agree to practice birth control and not donate sperm while on the study and for 3 months after, if a man. (This study has been changed. Male volunteers are now prohibited from donating sperm.)
* Have a stable weight during the past 6 months of at least 110 pounds and are close to ideal body weight.

Exclusion Criteria

Volunteers will not be eligible for this trial if they:

* Are women able to have children.
* Have heart or blood disease, kidney disease, stomach or intestinal problems, conditions affecting the nervous system, hormonal problems, any immune system problems, lung disease, or mental conditions, including the following: high blood pressure, heart disease, diabetes, asthma, elevated cholesterol, elevated triglycerides, inflamed pancreas, and blood-clotting disorders requiring anticoagulation.
* Have any stomach or intestinal problem that may interfere with the ability to take drugs
* Have any other medical condition that may interfere with being part of the study.
* Have been diagnosed with serious mental disorders such as depression, bipolar affective disorder, schizophrenia, or attempted suicide. Patients who have had less serious mental conditions that have been resolved may be included in the study, with approval.
* Have received protease inhibitors, nonnucleoside reverse transcriptase inhibitors, or experimental agents (not approved by the FDA for the use for which it is being tested) within 60 days of study entry.
* Have received treatment for an infection or other medical illness within 14 days of study entry.
* Have had high unexplained fever, or an illness with high fever lasting 3 or more days within 14 days of study entry.
* Have a history of allergies to any of the study drugs or their components, such as gelatin.
* Have used prescribed medications within 14 days of study entry.
* Have used natural or homeopathic remedies including herbal teas within 14 days of entering the study.
* Are unable to follow the schedule for study drugs during the trial.
* Are unable to participate in the blood level studies.
* Actively abuse drugs or alcohol.
* Change existing tobacco smoking habits during the study.
* Cannot avoid strenuous exercise or constant activity for the study period.
* Cannot avoid taking caffeine or alcohol at certain times before the blood level studies.
* Have had an allergic reaction to any drugs.
* (This protocol has been changed. Entry criteria are different from the original.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2001-03; Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gene Morse, Study Chair
Locations (8):
- United States (8):
  - Stanford CRS, Palo Alto, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - The Ohio State University Medical Center, Columbus, Ohio
  - Vanderbilt Univ. Med. Ctr., AIDS Clinical Trials Ctr., Nashville, Tennessee
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Result] Morse GD, Rosenkranz S, Para MF, Segal Y, Difrancesco R, Adams E, Brizz B, Yarasheski KE, Reichman RC. Amprenavir and efavirenz pharmacokinetics before and after the addition of nelfinavir, indinavir, ritonavir, or saquinavir in seronegative individuals. Antimicrob Agents Chemother. 2005 Aug;49(8):3373-81. doi: 10.1128/AAC.49.8.3373-3381.2005. PMID 16048950